CLINICAL TRIAL: NCT05621395
Title: A Randomized, Double-blind, Placebo-Controlled Study to Explore the Effect of E-OJ-01 on Fatigue and Cardiorespiratory Fitness in Healthy Adults.
Brief Title: To Study the Effect of Investigational Product on Fatigue and Cardiorespiratory Fitness in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EB/220604/OXY/FATIGUE
Record Dates: First submitted 2022-11-01; First posted 2022-11-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-OJ-01 (Experimental): 1 capsule (400 mg) orally to be taken after breakfast daily for 60 days
  Interventions: Other: E-OJ-01
- Microcrystalline cellulose (Placebo Comparator): 1 capsule (400 mg) orally to be taken after breakfast daily for 60 days
  Interventions: Other: Microcrystalline cellulose

INTERVENTIONS:
Other: E-OJ-01 — 1 capsule (400 mg) orally to be taken after breakfast daily for 60 days
  Arms: E-OJ-01
Other: Microcrystalline cellulose — 1 capsule (400 mg) orally to be taken after breakfast daily for 60 days
  Arms: Microcrystalline cellulose

SUMMARY:
E-OJ-01 (Oxyjun®), a proprietary, standardized aqueous extract of TA, has been proven to improve cardiac output and thereby lead to better oxygenation capacity and exercise endurance.

This, in turn, averts fatigue and improves physical functioning. Based on the previous studies of E-OJ-01 and the scientific literature available in support of the antioxidant and anti- inflammatory activity of TA bark, in the present study, it is hypothesized that E-OJ-01 will be able to reduce fatigue and improve the cardiorespiratory fitness of the male participants aged between 30 to 60 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males aged ≥30 to ≤60 years.
2. Body mass index (BMI) ≥18 and ≤29.9 kg/m2
3. VO2 max ≥20 ml/kg/ min but ≤35 ml /min/kg.
4. FAS total score ≥22.
5. Systolic blood pressure (SBP) ≤130 mm Hg and diastolic blood pressure (DBP) ≤89 mm Hg.
6. Ready to abstain from alcohol, caffeine, and vigorous physical activity for 24 h before every study visit.
7. Individuals who can comply and perform the procedures as per the protocol (consumption of study medications, biological sample collection procedures, and study visit schedule).
8. Individuals who are literate enough to understand the purpose of the study and their rights.
9. Individuals who can give written informed consent and are willing to participate in the study.

Exclusion Criteria:

1. Individuals with a history of any pulmonary disorder.
2. Known cases of hypertension and diabetes mellitus.
3. SpO2 < 96%
4. Random blood glucose (RBG) levels ≥140 mg/dl.
5. Hemoglobin (Hb) <13.0 g/dl.
6. Abnormal thyroid stimulating hormone (TSH) value (<0.4μIU/ml or >4.2μIU/ml).
7. Individuals with a history of COVID-19 in the last 3 months.
8. Individuals currently on/or having a history of taking blood lipid-lowering medications.
9. Individuals who are unable to run due to any joint disorder.
10. History of smoking or active smokers using any form of tobacco.
11. Individuals with substance abuse problems (within two years) defined as:

    * Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
    * High-risk drinking as defined as consuming 5 or more alcohol-containing drinks on any day or 15 or more alcohol-containing drinks per week.
12. Individuals who are currently on dietary supplements.
13. Individuals who are currently on diuretics.
14. History/symptoms of any cardiovascular disorder such as coronary artery disease or myocardial infarction.
15. Individuals having clinically significant illnesses of the endocrine, immune, gastrointestinal, hepatobiliary, kidney, urinary, hematological, musculoskeletal system, and/or any inflammatory disorder.
16. History of any significant neurological and psychiatric condition, which may affect the participation and inference of the studys endpoints.
17. Participation in other clinical trials in the last 90 days before screening.
18. Any condition that could, in the opinion of the Investigator, preclude the participants ability to successfully and safely complete the study or may confound study outcomes.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Day 0 baseline to Day 60
  To determine the effect of 60 days of product on exercise capacity as assessed by change in time-to-exhaustion (TTE) as evaluated by the Borg RPE scale while running on a treadmill using the Modified Bruce treadmill test protocol compared to the placebo. It is a 15-point single-item scale ranging from 6 to 20, with anchors ranging from 6 "No exertion" to 20 "Maximum exertion"The Borg Score of ≥ 19 will indicate the point of volitional exhaustion, and the exercise protocol will be terminated at this point.

SECONDARY OUTCOMES:
Cardiorepiratory fitness | Day 0 and Day 60
  The most accurate assessment of VO2 max is made by measuring expired air composition and respiratory volume during maximal exertion. VO2 max can be estimated from the peak exercise intensity during a maximal exercise test. The primary criterion for attaining VO2 max is a plateau in VO2. Several secondary criteria exist in the case of a plateau in VO2 not being reached, which include a rise in respiratory exchange ratio above 1.0 depending on the age, blood lactate concentration above 8 mmol/l, and an increase in heart rate to the age-predicted maximum.
Exercise-induced fatigue and energy levels | Day 0 and Day 60
  The Visual Analog Scale for energy is anchored with the verbal cues "low" and "high", while VAFS is anchored with the verbal cues "no fatigue" and "very severe fatigue". A higher score indicates higher energy and fatigue on the respective scales
General fatigue | Day 0, Day 15, Day 30 and Day 60
  The scale score is calculated by summing all items. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest. A total FAS score < 22 indicates no fatigue, and a score ≥ 22 indicates fatigue.The Minimal Clinically Important Difference (MCID) of at least 4 points or 10% change of the baseline value has been reported in cases of sarcoidosis.
Physical fatigue | Day 0, Day 15, Day 30 and Day 60
  The scale score is calculated by summing all items. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest. A total FAS score < 22 indicates no fatigue, and a score ≥ 22 indicates fatigue.The Minimal Clinically Important Difference (MCID) of at least 4 points or 10% change of the baseline value has been reported in cases of sarcoidosis.
Heart rate at maximal fatigue | Day 0 and Day 60
  Higher the percentile superior is the health
Mitochondrial biogenesis | Day 0 and Day 60
  Energy balance as assessed by serum PGC-1α levels, a marker of mitochondrial biogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Study Director — Vedic Lifesciences Pvt. Ltd.
Locations (4):
- India (4):
  - D.Y. Patil deemed to be University,, Nerul, Maharashtra
  - Dr. Preeti Bawaskar's Clinic, Thane, Maharashtra
  - Shree Ashirwad Hospital, Thane, Maharashtra
  - Jaipur National University Institute for Medical Science and Research Centre, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided